CLINICAL TRIAL: NCT01851590
Title: Efficacy of Topical Resin Lacquer, Amorolfine, and Oral Terbinafine for Treating Toenail Onychomycosis: a Prospective, Randomized, Controlled, Investigator-blinded, Parallel-group Clinical Trial
Brief Title: Resin vs. Amorolfine vs. Terbinafine Treatment in Onychomycosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Repolar Pharmaceuticals Oy (Industry)
Responsible Party: Principal Investigator, Janne J. Jokinen, Consultant Cardiothoracic Surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 334/13/03/01/2012; 2012-004822-48 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Onychomycosis
Keywords: Dermatophyte onychomycosis; Fungal nail infection; Resin Lacquer; Amorolfine; Terbinafine
MeSH Terms: conditions — Onychomycosis | interventions — amorolfine; Terbinafine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resin Lacquer (Experimental): Topical 30% Resin Lacquer applied once daily for 9 months (Abicin® 30% Nail Lacquer).
  Interventions: Device: Resin Lacquer
- Amorolfine (Active Comparator): Topical 5% Amorolfine Lacquer applied once weekly for 9 months (Loceryl® 5% Nail Lacquer).
  Interventions: Drug: Amorolfine
- Terbinafine (Active Comparator): 250 mg of Terbinafine taken orally once daily for 3 months (Generics).
  Interventions: Drug: Terbinafine

INTERVENTIONS:
Device: Resin Lacquer — 30% Resin Lacquer is applied once daily for 9 months (Abicin®) in toenail onychomycosis.
  Other Names: Resin Lacquer arm
  Arms: Resin Lacquer
Drug: Amorolfine — 5% Amorolfine Lacquer is applied once weekly for 9 months (Loceryl®) in toenail onychomycosis.
  Other Names: Amorolfine Lacquer arm
  Arms: Amorolfine
Drug: Terbinafine — 250 mg of Terbinafine is taken orally once daily for 3 months (Generics) in toenail onychomycosis.
  Other Names: Terbinafine arm
  Arms: Terbinafine

SUMMARY:
The current study is conducted to corroborate the previous observational clinical trial with more valid methods and a more clinically relevant experimental design. This study aims to compare efficacy, safety, and cost between topically administered 30% resin lacquer for the treatment of dermatophyte toenail onychomycosis and the current "best practices": topical 5% amorolfine and systemic terbinafine.

DETAILED DESCRIPTION:
The aim of this prospective, investigator-blinded, randomized and controlled clinical trial is to explore potential differences between 5 % amorolfine and 30 % resin lacquer in topical treatment of onychomycosis. In addition, topical treatment methods are compared with the most effective 'drug of choice' for onychomycosis according the current guidelines i.e. oral medication with terbinafine.

Altogether 90 patients (the aim is to collect the 30 patients per group) who have culture or potassium hydroxide (KOH) stain verified dermatophyte onychomycosis are randomly allocated into 3 treatment groups to receive either topical treatment or oral medication for toenail onychomycosis classified as follows:

1. White superficial onychomycosis (WSO)
2. Distal and lateral subungual onychomycosis (DLSO)
3. Proximal subungual onychomycosis (PSO)
4. [Total dystrophic onychomycosis) (TDO)] [Excluded]
5. [Candidal onychomycosis] [Excluded]

Participants are randomized into 3 groups to receive:

1. Topical treatment: 30 % resin lacquer (Abicin®) applied once daily for 9 months.
2. Topical treatment: 5 % amorolfine lacquer (Loceryl®) applied once weekly for 9 months.
3. Oral medication: 250 mg terbinafine taken orally once daily for 3 months.

All patients visit at outpatient department before the launch of the study, and 3 and 9 months thereafter. Clinical examination is done by 4 physicians. During the 42-week study period, laboratory tests are conducted on samples collected before treatment, at 20 weeks, and at 42 weeks. The tests include a fungal culture, KOH staining of the toenail sample, and blood tests. Cultures and KOH microscopy are performed in an independent, specialised mycology laboratory with standard techniques (Medix Laboratories Ltd., Helsinki, Finland). The blood tests measure plasma γ-glutamyl transferase levels (also at 2 weeks); plasma creatinine levels; the total number of white blood cells, including neutrophils, monocytes, basophils, lymphocytes, and eosinophils; the total number of red blood cells, including erythrocytes and haematocrit; erythrocyte indices, including the mean corpuscular volume, mean corpuscular haemoglobin, mean corpuscular haemoglobin concentration, and haemoglobin level; and the total number thrombocytes (initially and at 42 weeks). During the control visits, sequential digital photographs of the most disfigured and brittle toenails are acquired.

In the three phone calls, patients are asked about potential treatment-related side effects, compliance with treatment, patients' perception of treatment outcome, and their willingness to continue in the study. In each treatment arm, the treatment regimen is discontinued 5 weeks before the last toenail sampling to provide an appropriate washout period before the final culture and KOH analysis.

To ensure safety and to assess potential contraindications for the treatment regimens, all patients included in the study undergo a comprehensive medical interview and physical examination. To identify patients who may develop intolerable adverse events due to drug combinations, all concurrent medications are cross-checked to verify compatibility with resin, amorolfine, and terbinafine regimens at the beginning of the study. All patients are informed of the possibility of developing a hypersensitivity to resin, amorolfine, or terbinafine. If patients experienced symptoms that corresponded to any level of hypersensitivity, they are dropped from the study.

ELIGIBILITY:
Inclusion Criteria:

* Positive dermatophyte culture in the beginning of the study obtained from the toenail sample.
* Positive KOH stain in the beginning of the study obtained from the toenail sample.

Exclusion Criteria:

* Any other nail disease than dermatophyte culture or KOH stain verified onychomycosis
* Onychomycosis caused by yeasts or nondermatophyte molds
* Kidney failure determined by plasma creatinine level (P-Krea > 100 μmol/l)
* Liver failure determined by plasma γ-glutamyltransferase level (P-GT > 120 U/I)
* Sensitivity or allergy to Resin, Amorolfine or Terbinafine
* Potential adverse cross-reaction of Terbinafine, Amorolfine or Resin with the patient's permanent medication
* Presence of total dystrophic onychomycosis (TDO)
* Any topical or oral antifungal treatment within the 6 months before the beginning of the study (washout period > 6 months).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janne J. Jokinen, MD, PhD, Principal Investigator — Department of Cardiac Surgery, Heart and Lung Centre, Helsinki University Hospital, FI-00029, Helsinki, Finland
Locations (2):
- Finland (2):
  - Vääksyn Lääkärikeskus, Vääksy, Vääksy
  - Vääksyn Lääkärikeskus, Vääksy

REFERENCES:
- [Background] Sigurgeirsson B et al. Efficacy of amorfine nail lacquer for the prophylaxis of onychomycosis over 3 years. J Eur Acad Dermatol Venereol 2010;24: 910-5. Rautio M et al. Antibacterial effects of home-made resin salve from Norway spruce (Picea abies). APMIS 2007;115: 335-340. Rautio M et al. In vitro fungistatic effects of natural coniferous rosin from Norway spruce (Picea abies). Eur J Clin Microbiol Infect Dis 2012;31:1783-9. Sipponen A et al. Effects of Norway spruce (Picea abies) resin on cell wall and cell membrane of Staphylococcus aureus. Ultrastruct Pathol 2009;33: 128-135. Sipponen P et al. Natural coniferous resin lacquer in treatment of toenail onychomycosis: an observational study. Mycoses 2012, Accepted. Roberts DT et al. British Association of Dermatologists. Guidelines for treatment of onychomycosis. Br J Dermatol 2003;148:402-10. Baran R et al. A new classification of onychomycosis. Br J Dermatol 1998;139: 567-71.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In November 2013, on the basis of a newspaper advertisement, a total of 129 adult volunteers were assessed for eligibility at Vääksy Medical Center, Finland. Eligible subjects were required to provide toenail samples for screening. Inclusion criteria were a positive dermatophyte culture and a positive potassium hydroxide (KOH) stain.
Pre-assignment Details: Of those 129 patients screened, 48 (37%) were excluded due to negative KOH staining or cultures and 8 (6%) were excluded because onychomycosis was caused by nondermatophyte mold or yeast. At baseline, 73 (57%) patients who met the entry criteria were randomly allocated to receive 1 of 3 therapies for dermatophyte onychomycosis (3 treatment arms).
Groups:
- Resin Lacquer Arm: Topical treatment: 30 % Resin Lacquer (Abicin®)
  Resin Lacquer was administered locally in the form of lacquer (Abicin®) onto infected nail once a day for 9 months in toenail onychomycosis.
- Amorolfine Lacquer Arm: Topical treatment with 5 % Amorolfine Lacquer (Loceryl®)
  Amorolfine: Amorolfine was administered locally in the form of lacquer (Loceryl®) onto infected nail once a week for 9 months in toenail onychomycosis.
- Terbinafine Arm: Oral medication with 250 mg terbinafine / day
  Terbinafine: Terbinafine 250 mg was administered orally once a day for 3 months in toenail onychomycosis.
Period: Overall Study
Arm/Group | Resin Lacquer Arm | Amorolfine Lacquer Arm | Terbinafine Arm
Started | 23 (In addition to clinical control visits, patients were contacted by phone during weeks 6, 13, and 29.) | 25 (In addition to clinical control visits, patients were contacted by phone during weeks 6, 13, and 29.) | 25 (In addition to clinical control visits, patients were contacted by phone during weeks 6, 13, and 29.)
At 3 Month: End of Terbinafine Treatment | 23 (Topical Resin Lacquer treatment continues ->) | 24 (Topical Amorolfine Lacquer Treatment continues ->) | 22 (End of oral Terbinafine treatment. Washout period of the Terbinafine treatment arm begins.)
At 4 Month: Follow-up Visit and Control | 23 (Clinical response to treatment, toenails samples and laboratory exams were controlled.) | 24 (Clinical response to treatment, toenails samples and laboratory exams were controlled.) | 22 (Clinical response to treatment, toenails samples and laboratory exams were controlled.)
At 9 Month: End of Topical Treatments | 23 (End of topical Resin Lacquer treatment. Washout period of the Resin Lacquer treatment arm begins.) | 24 (End of topical Amorolfine Lacquer treatment. Washout period of the Amorolfine treatment arm begins.) | 22 (Washout period of the Terbinafine treatment arm continues.)
At 10 Month: Follow-up Visit and Control | 23 (Study completed. Clinical response to treatment, toenails samples and lab. exams were controlled.) | 24 (Study completed. Clinical response to treatment, toenails samples and lab. exams were controlled.) | 22 (Study completed. Clinical response to treatment, toenails samples and lab. exams were controlled.)
Completed | 23 (All patients (23) were included in the ITT population and final outcome analyses.) | 24 (All patients (25) were included in the ITT population and final outcome analyses.) | 22 (All patients (25) were included in the ITT population and final outcome analyses.)
Not Completed | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Primary and secondary outcome analyses were based on the intent-to-treat (ITT) population and missing values were imputed using the last observation carried forward (LOCF) method. At baseline, 73 patients who met the entry criteria were randomized to one of the three arms: topical Resin Lacquer, topical Amorolfine Lacquer or oral Terbinafine.
Groups:
- Resin Lacquer Arm: Topical treatment: 30 % Resin Lacquer (Abicin®)
  Resin Lacquer is administered locally in the form of lacquer (Abicin®) onto infected nail once a day for 9 months in toenail onychomycosis.
- Amorolfine Lacquer Arm: Topical treatment with 5 % Amorolfine Lacquer (Loceryl®)
  Amorolfine Lacquer is administered locally in the form of lacquer (Loceryl®) onto infected nail once a week for 9 months in toenail onychomycosis.
- Terbinafine Arm: Oral medication with 250 mg Terbinafine / day
  Terbinafine 250 mg is administered orally once a day for 3 months in toenail onychomycosis.
- Total: Total of all reporting groups
Arm/Group | Resin Lacquer Arm | Amorolfine Lacquer Arm | Terbinafine Arm | Total
Number analyzed (Participants) | 23 | 25 | 25 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 20 | 58
  >=65 years | 5 | 5 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 8 | 15
  Male | 21 | 20 | 17 | 58
Region of Enrollment [Number; unit: participants]
  Finland | 23 | 25 | 25 | 73
Positive mycological culture in toenail samples [Number; unit: participants] | 23 | 25 | 25 | 73
BMI [Mean (Standard Deviation); unit: kg/m^2] — kg/m2
  kg/m^2 | 25 (3) | 27 (4) | 27 (4) | 26 (4)
Specific dermatophyte species in mycological culture [Number; unit: participants]
  Trichophyton rubrum | 20 | 24 | 21 | 65
  Trichophyton mentagrophytes | 3 | 1 | 4 | 8
Plasma creatinine [Mean (Standard Deviation); unit: μmol/l] | 76 (15) | 78 (13) | 79 (11) | 78 (14)
Plasma γ-glutamyl transferase [Median (Inter-Quartile Range); unit: U/I] | 29 [17 to 41] | 21 [14 to 41] | 27 [18 to 47] | 25 [20 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Mycological Cure
Description: To analyze the rate of complete mycological cure i.e. fungal eradication in terms of negative mycological culture AND negative potassium hydroxide (KOH) stain at 4- and 10 months time-points from the beginning of the study.
Time Frame: At 4- and 10 months time-points from the beginning of the study.
Population: Primary and secondary outcome analyses were based on the intent-to-treat (ITT) population and missing values were imputed using the last observation carried forward (LOCF) method.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Resin Lacquer Arm: Topical treatment with 30 % Resin Lacquer (Abicin®)
  Resin is administered locally in the form of lacquer (Abicin®) onto infected nail once a day for 9 months in toenail onychomycosis.
- Amorolfine Lacquer Arm: Topical treatment with 5 % Amorolfine Lacquer (Loceryl®)
  Amorolfine is administered locally in the form of lacquer (Loceryl®) onto infected nail once a week for 9 months in toenail onychomycosis.
Arm/Group | Resin Lacquer Arm | Amorolfine Lacquer Arm | Terbinafine Arm
Number analyzed (Participants) | 23 | 25 | 25
Percentage of participants
  Mycological cure at 4-month | 17 [1 to 34] | 28 [9 to 47] | 16 [0 to 31]
  Mycological cure at 10-month | 13 [0 to 28] | 8 [0 to 19] | 56 [35 to 77]
Statistical Analysis 1: Comparison: Resin Lacquer Arm vs Amorolfine Lacquer Arm vs Terbinafine Arm; The sample size was estimated according to complete mycological cure at 10 months. Estimation was based on the design of a binary-outcome head-to-head superiority trial. Orally administered terbinafine treatment was considered the active control. Approximately 25 patients / arm were required to have 80% power (β=0.2) at a two-sided α=0.05 significance level to detect a decrease in primary outcome from 50% in the terbinafine arm to 15% in the amorolfine or resin lacquer treatment arms; Test type: Superiority or Other; p < 0.05, Cochran-Mantel-Haenszel — Proportions and 95% confidence intervals (CIs) were calculated for negative KOH staining, negative cultures, and a combination of these at 4- and 10-month time points. Cochran-Mantel-Haenszel and χ2-tests were used to analyse efficacy criteria

2. Secondary Outcome: Clinical Responses to the Treatments
Description: Clinical responses to treatment were based on the proximal linear growth of healthy nail; thus, the clinical responses were classified as partial (evident proximal linear growth of healthy nail) or complete. Partial responses were defined as significant reductions in onycholysis, subungual hyperkeratosis, and streaks. A complete response was a fully normal appearance of the toenail.
Time Frame: At 4- and 10 months time-points from the beginning of the study.
Population: Intention-to-treat population, last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Resin Lacquer Arm | Amorolfine Lacquer Arm | Terbinafine Arm
Number analyzed (Participants) | 23 | 25 | 25
percentage of participants
  Partial clinical response at 4-month | 0 | 0 | 44
  Complete clinical response at 4-month | 0 | 0 | 0
  Partial clinical response at 10-month | 30 | 28 | 36
  Complete clinical response at 10-month | 0 | 0 | 16
Statistical Analysis 1: Comparison: Resin Lacquer Arm vs Amorolfine Lacquer Arm vs Terbinafine Arm; Test type: Superiority or Other; p < 0.05, ANOVA — Differences between quantitative data were assessed with one-way analysis of variances, and pairwise comparisons were performed with Bonferroni's post hoc test

3. Secondary Outcome: Cost-effectiveness 1
Description: Cost analysis was based on the retail price (€) and consumption of a 10 ml bottle of Abicin® 30% resin lacquer, a 5 ml bottle of Loceryl® 5% amorolfine lacquer, and 98 tablets of generic 250 mg terbinafine, sold by the University Pharmacy in Helsinki, Finland, January 2014. The cost was expressed as the average treatment cost per patient; for the total cost, this average was extrapolated to the entire study treatment arm. The results show the treatment costs (€) per day per patient in each group.
Time Frame: At 10-month time-point
Measure: Mean (95% Confidence Interval); unit: Euros (€)
Groups:
- Amorolfine Treatment Arm: Topical treatment with 5 % amorolfine lacquer (Loceryl®)
  Amorolfine is administered locally in the form of lacquer (Loceryl®) onto infected nail once a week for 9 months in toenail onychomycosis.
Arm/Group | Resin Lacquer Arm | Amorolfine Treatment Arm | Terbinafine Arm
Number analyzed (Participants) | 23 | 25 | 25
Euros (€) | 0.15 [0.14 to 0.15] | 0.21 [0.20 to 0.21] | 0.56 [0.52 to 0.59]
Statistical Analysis 1: Comparison: Resin Lacquer Arm vs Amorolfine Treatment Arm vs Terbinafine Arm; Test type: Superiority or Other; p < 0.05, ANOVA — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Cost-effectiveness 2
Description: Cost analysis was based on the retail price (€) and consumption of a 10 ml bottle of Abicin® 30% resin lacquer, a 5 ml bottle of Loceryl® 5% amorolfine lacquer, and 98 tablets of generic 250 mg terbinafine, sold by the University Pharmacy in Helsinki, Finland, January 2014. The cost was expressed as the average treatment cost per patient; for the total cost, this average was extrapolated to the entire study treatment arm. The results show the treatment costs (€) during the treatment period per patient in each group.
Time Frame: At 10-month time-point
Measure: Mean (95% Confidence Interval); unit: Euros (€)
Arm/Group | Resin Lacquer Arm | Amorolfine Treatment Arm | Terbinafine Arm
Number analyzed (Participants) | 23 | 25 | 25
Euros (€) | 40.7 [38.8 to 42.6] | 55.2 [52.9 to 57.5] | 52.1 [46.8 to 53.0]
Statistical Analysis 1: Comparison: Resin Lacquer Arm vs Amorolfine Treatment Arm vs Terbinafine Arm; Test type: Superiority or Other; p < 0.05, ANOVA — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Compliance to the Treatment
Description: Evaluation of compliance was based on patient self-reports of whether the treatment protocol was followed 100% (complete), 80% (good), 60% (moderate), or 40% (poor) of the time.
Time Frame: At 4-month time-point
Population: Percentage describes the proportion of patients who declared that they have been followed the instructions completely (100%).
Measure: Number; unit: percentage of participants
Arm/Group | Resin Lacquer Arm | Amorolfine Lacquer Arm | Terbinafine Arm
Number analyzed (Participants) | 23 | 25 | 25
percentage of participants | 100 | 96 | 100
Statistical Analysis 1: Comparison: Resin Lacquer Arm vs Amorolfine Lacquer Arm vs Terbinafine Arm; Test type: Superiority or Other; p < 0.05, Chi-squared — Qualitative data are expressed as frequencies and percentages, and differences between parallel groups were compared with the χ2-test or Fisher's exact test, as appropriate

ADVERSE EVENTS:
Time Frame: Adverse effects or side-effects during the 10-month follow-up
Description: All side-effects or adverse events were recorded systematically. Information on the side-effects were specifically asked by the research coordinator during the two follow-up visits (at 4- and 10-month) and three telephone contacts. Patients were asked to contact research coordinator if any obvious or suspected side-effect would emerge.
Arm/Group | Resin Lacquer Arm | Amorolfine Lacquer Arm | Terbinafine Arm
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resin Lacquer Arm (N=23) | Amorolfine Lacquer Arm (N=25) | Terbinafine Arm (N=25)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
* Relatively short treatment period for the toenail onychomycosis (9 months).
* Patients with total dystrophic onychomycosis (46%) - the most difficult subtype to treat - may not have been amenable to monotherapy with a topical antifungal treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No